CLINICAL TRIAL: NCT04314960
Title: Immediate and Long-term Effects of Gait Training With Functional Electrical Stimulation in Subjects With Chronic Ankle Instability
Brief Title: Functional Electrical Stimulation in Chronic Ankle Instability
Acronym: ESCAIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shmuel Springer (Other)
Responsible Party: Sponsor-Investigator, Shmuel Springer, Chair, Physiotherapy Department, Neuromuscular & Human Performance Laboratory, Ariel University
Organization: Ariel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU-HEA-SS-20200308a
Record Dates: First submitted 2020-03-15; First posted 2020-03-19 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Joint Instability; Ankle Sprains; Sport Injury
Keywords: Chronic ankle instability; Rehabilitation; Neuromuscular control; Gait; Electrical stimulation
MeSH Terms: conditions — Joint Instability; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CAI subjects (Experimental): Subjects in this group will receive eight 20-minutes gait training sessions with functional electrical stimulation.
  Interventions: Device: Functional electrical stimulation device (NESS L300Plus, Bioness, Valencia, CA)

INTERVENTIONS:
Device: Functional electrical stimulation device (NESS L300Plus, Bioness, Valencia, CA) — Functional electrical stimulation (FES) is the application of high-intensity intermittent electrical stimuli to generate muscle contractions that may bypass spinal and supraspinal inhibition, and which is coupled with a functional task such as gait. Gait training will be conducted on a treadmill.

SUMMARY:
Individuals with chronic ankle instability (CAI) display neuromuscular deficits such as altered control of posture and gait when compared with healthy controls. These deficits may be attributed to muscle inhibition occurring after a surrounding joint structure has been damaged. Functional electrical stimulation (FES) is the application of high-intensity intermittent electrical stimuli to generate muscle contractions that may overcome inhibition, and which is coupled with a functional task such as gait.

The current study aims to investigate the short and immediate effects of FES on gait parameters and postural control in subjects with CAI. Prior to intervention, treadmill gait will be evaluated using a motion analysis system, and postural control will be evaluated in a series of tests that measure balance, reaction time to ankle perturbation and stabilization ability after jump-landing. Then, a 20 minutes gait training with an FES device will be applied. Immediate effects of the training on gait parameters will be assessed. For medium-term effects evaluation, subjects will return for additional 7 training sessions (2 per week for 4 weeks), following by a complete measurements acquisition as prior to intervention. At six months follow-up, subjects will be contacted for collecting subjective outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. A history of at least one significant ankle sprain:

   1. At least 12 months prior to participating in the study
   2. Was characterized by inflammatory symptoms (i.e. pain and swelling)
   3. Caused at least one day of decreased physical activity
2. At least 3 months since the last acute ankle sprain that results in inflammatory symptoms and at least one interrupted day of desired physical activity.
3. History of the previously injured ankle 'giving way' at least twice during the last 6 months, and/or 'feelings of instability' and/or recurrent sprain.
4. Being able to bear full weight on the injured lower extremity with no more than mild discomfort.
5. Scoring<24 in the Cumberland Ankle Instability Tool (CAIT)

Exclusion Criteria:

1. A history of previous surgeries to a musculoskeletal structure in either lower limb.
2. A history of a fracture requiring re-alignment
3. Any acute injury to a lower limb in the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Immediate change in ankle inversion angle during heel strike | immediately after the intervention
  Ankle inversion angle at heel strike (in degrees) will be measured using Qualisys motion analysis system.
  Change will be measured between pre-intervention to immediately after first intervention session to assess immediate effects of the intervention.
Change in ankle inversion angle during heel strike at 4 weeks | through intervention completion, approximately at 4 weeks
  Ankle inversion angle at heel strike (in degrees) will be measured using Qualisys motion analysis system.
  Change will be measured between pre-intervention and after completing the entire intervention.
Immediate change in peroneal muscle electromyography | immediately after the intervention
  Peroneal muscle activity will be measured (in millivolts) using Trigno EMG system during the 5% of gait cycle prior to heel strike.
  Change will be measured between pre-intervention to immediately after first intervention session to assess immediate effects of the intervention.
Change in peroneal muscle electromyography at 4 weeks | through intervention completion, approximately at 4 weeks
  Peroneal muscle activity will be measured (in millivolts) using Trigno EMG system during the 5% of gait cycle prior to heel strike.
  Change will be measured between pre-intervention and after completing the entire intervention.

SECONDARY OUTCOMES:
Change in Star excursion balance test (SEBT) score | through intervention completion, approximately at 4 weeks
  The SEBT has been previously described as a postural control test that can differ between subjects with CAI and healthy controls. The test is performed with the subjects standing barefoot in the middle of a grid formed by eight tape measures extending out at 45° from each other. While the subject is balancing on one leg that is placed in the middle of the grid, the other leg has to reach as far as possible in each direction. The reached distance in centimeters is recorded, with the greater distance representing better postural stability. An average scores is calculated and normalized to the length of the subject's leg in centimeters.
Time to stabilization (TTS) | through intervention completion, approximately at 4 weeks
  TTS is the time required to normalize ground reaction forces (GRF) after following a jump-landing. To measure TTS, subjects will be required to perform a single-leg drop-jump from a 40-cm box onto a force plate (Kistler, Switzerland) and keep balancing on a single leg for 20 seconds. GRF recordings will be analyzed to determine TTS in seconds in the ML and AP planes, as was previously described. Shorter duration demonstrates better postural stability. Subjects will be allowed at least 3 practice trials, following by 5 successful jumps landings. A rest period of 30 seconds will be allowed between jumps. If a subject will not be able to stabilize for at least 20 seconds, the trial will be repeated.
  Lower values indicate better postural control.
Peroneal reaction time (PRT) | through intervention completion, approximately at 4 weeks
  PRT is the time duration between and ankle inversion perturbation and beginning of peroneal muscle activation which is recognized using EMG. Subjects will stand on an inversion stimulator. In an unknown time, a sudden inversion perturbation will occur. Time measurement between perturbation time and muscle activation time is measured in seconds.
  Lower values indicate better postural control.

OTHER OUTCOMES:
Foot and Ankle Ability Measure (FAAM) - questionnaire | through intervention completion, approximately at 4 weeks
  A self-reported functional outcome measure utilized to track subjective changes in perceived pain and ankle function
  Score ranges between 0-100. Higher scores represent higher levels of function, with score of 100 represents no disability.
Cumberland Ankle Instability Tool (CAIT) - questionnaire | through intervention completion, approximately at 4 weeks
  A self-reported outcome measure designated for people with chronic ankle instability. Will also serve as an inclusion criteria.
  Score ranges between 0-30, with lower scores indicate less ankle instability.

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Springer, PhD, Principal Investigator — Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
Not decided yet, but optional to share all data after concealing subject's identifying details.